CLINICAL TRIAL: NCT05478382
Title: Efficacy and Side Effect Profile of Varying Dose of Pregabalin for the Treatment of Acute Postoperative Pain Following Spinal Surgery
Brief Title: Pregabalin is an Effective Treatment for Acute Postoperative Pain Following Spinal Surgery Without Major Side Effects
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ajou University School of Medicine (Other)
Collaborators: HK inno.N Corporation (Industry)
Responsible Party: Principal Investigator, Han Dong Lee, Assistant Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KAB 1.0
Record Dates: First submitted 2022-06-06; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Postoperative Pain; Pregabalin; Spine Surgery; Adverse Reaction to Pregabalin
Keywords: Postoperative Pain; pregabalin; Spine surgery; adverse reaction to pregabalin
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): 3 capsules of placebo drug are administered once prior to surgery and every 12 hours after surgery for 72 hours
  Interventions: Drug: Placebo
- Pregabalin 25mg (Experimental): 1 capsule of Kabalin 25mg Cap and 2 pills of placebo drug are administered once prior to surgery and every 12 hours after surgery for 72 hours
  Interventions: Drug: Pregabalin 25 MG; Drug: Placebo
- Pregabalin 50mg (Experimental): 2 capsules of Kabalin 25mg Cap and 1 pill of placebo drug are administered once prior to surgery and every 12 hours after surgery for 72 hours
  Interventions: Drug: Pregabalin 25 MG; Drug: Placebo
- Pregabalin 75mg (Experimental): 3 capsules of Kabalin 25mg Cap are administered once prior to surgery and every 12 hours after surgery for 72 hours
  Interventions: Drug: Pregabalin 25 MG

INTERVENTIONS:
Drug: Pregabalin 25 MG — Patients are given 0 to 3 capsules per administration according to their allocated group.
  Arms: Pregabalin 25mg; Pregabalin 50mg; Pregabalin 75mg
Drug: Placebo — Patients are given 0 to 3 capsules per administration according to their allocated group.
  Arms: Placebo; Pregabalin 25mg; Pregabalin 50mg

SUMMARY:
The objective of this study is to examine the efficacy and side effect of varying dose of pregabalin for the treatment of postoperative pain after spinal surgery.

DETAILED DESCRIPTION:
Patients experience considerable postoperative pain after spine surgery. Because the spine is located at the center of the body and supports body weight, severe postoperative pain hinders upper body elevation and gait which can lead to various complications such as pulmonary deterioration or pressure sores. It is important to effectively control postoperative pain to prevent such complications. Gabanoids are widely used as preemptive multimodal analgesia while their effects and side effects are known to be dose dependent. The objective of this study is to examine the efficacy and side effect of varying dose of pregabalin for the treatment of postoperative pain after spinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient undergoing spine surgery at out institution for degenerative lumbar disorder.

Exclusion Criteria:

* ASA classification over 2
* Patients with dizziness or frequent headache
* Active alcohol or drug usage
* Intake of any analgesics daily or 48 hours before surgery
* Impaired renal and/or hepatic function
* Diagnosed and being treated for anxiety or depression disorders
* Coverage from worker's compensation insurance or car insurance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Arrival at the general ward
  Change of Visual analogue scale (VAS) pain score
Pain intensity | 6hours after surgery
  Change of Visual analogue scale (VAS) pain score
Pain intensity | 24hours after surgery
  Change of Visual analogue scale (VAS) pain score
Pain intensity | 48hours after surgery
  Change of Visual analogue scale (VAS) pain score
Pain intensity | 72hours after surgery
  Change of Visual analogue scale (VAS) pain score
IV PCA usage | Arrival at the general ward
  amount of infused fentanyl-based intravenous patient-controlled analgesia (PCA)
IV PCA usage | 6hours after surgery
  amount of infused fentanyl-based intravenous patient-controlled analgesia (PCA)
IV PCA usage | 24hours after surgery
  amount of infused fentanyl-based intravenous patient-controlled analgesia (PCA)
IV PCA usage | 48hours after surgery
  amount of infused fentanyl-based intravenous patient-controlled analgesia (PCA)
IV PCA usage | 72hours after surgery
  amount of infused fentanyl-based intravenous patient-controlled analgesia (PCA)
Rescue analgesic usage | Arrival at the general ward
  Frequency of rescue analgesic administered
Rescue analgesic usage | 6hours after surgery
  Frequency of rescue analgesic administered
Rescue analgesic usage | 24hours after surgery
  Frequency of rescue analgesic administered
Rescue analgesic usage | 48hours after surgery
  Frequency of rescue analgesic administered
Rescue analgesic usage | 72hours after surgery
  Frequency of rescue analgesic administered

SECONDARY OUTCOMES:
Nausea and vomiting due to IV PCA usage | From arrival at general ward after sugery for 72 hours, subdivided into 4 periods (1-6hours, 6-24hours, 24-48hours, 48-72hours)
  Incidence and frequency of nausea and vomiting event due to IV PCA usage

CONTACTS AND LOCATIONS:
Overall Officials: Han-Dong Lee, Prof., Principal Investigator — Ajou University Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Helenius L, Yrjala T, Oksanen H, Pajulo O, Loyttyniemi E, Taittonen M, Helenius I. Pregabalin and Persistent Postoperative Pain Following Posterior Spinal Fusion in Children and Adolescents: A Randomized Clinical Trial. J Bone Joint Surg Am. 2021 Dec 1;103(23):2200-2206. doi: 10.2106/JBJS.21.00153. Epub 2021 Aug 23. PMID 34424869
- [Background] Helenius LL, Oksanen H, Lastikka M, Pajulo O, Loyttyniemi E, Manner T, Helenius IJ. Preemptive Pregabalin in Children and Adolescents Undergoing Posterior Instrumented Spinal Fusion: A Double-Blinded, Placebo-Controlled, Randomized Clinical Trial. J Bone Joint Surg Am. 2020 Feb 5;102(3):205-212. doi: 10.2106/JBJS.19.00650. PMID 31770296
- [Background] Kim JC, Choi YS, Kim KN, Shim JK, Lee JY, Kwak YL. Effective dose of peri-operative oral pregabalin as an adjunct to multimodal analgesic regimen in lumbar spinal fusion surgery. Spine (Phila Pa 1976). 2011 Mar 15;36(6):428-33. doi: 10.1097/BRS.0b013e3181d26708. PMID 21372654
- [Background] Panse NA, Adate KU, Panchal SH. Comparative Evaluation of Two Different Doses of Pre-Emptive Oral Pregabalin on Duration of Spinal Anesthesia and Postoperative Pain. Archives of Anesthesiology and Critical Care. 2021;7(2):75-81
- [Derived] Park KH, Chung NS, Chung HW, Kim TY, Lee HD. Pregabalin as an effective treatment for acute postoperative pain following spinal surgery without major side effects: protocol for a prospective, randomized controlled, double-blinded trial. Trials. 2023 Jun 22;24(1):422. doi: 10.1186/s13063-023-07438-2. PMID 37349841